CLINICAL TRIAL: NCT03160287
Title: Mobile Motivational Physical Activity Targeted Intervention (MobMPATI) to Improve Sleep in Older Adults With Osteoarthritis
Brief Title: Mobile Motivational Physical Activity Targeted Intervention
Acronym: MobMPATI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Oleg Zaslavsky, Assistant Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 52062
Record Dates: First submitted 2017-04-20; First posted 2017-05-19 (Actual); Results first posted 2021-05-21 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Osteoarthritis
Keywords: mobile, sleep, physical activity, older adults
MeSH Terms: conditions — Osteoarthritis; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Motivational interview and text messages (Experimental): Multidimensional, tailored intervention for sleep deficiency in for older adults with OA
  Interventions: Behavioral: Motivaltional interviews and infrequent motivational text messages

INTERVENTIONS:
Behavioral: Motivaltional interviews and infrequent motivational text messages — A self-management intervention will integrate use of mobile technology to prompt older adults to be physically active, provides ongoing monitoring of the amount of their physical activity and includes self-efficacy enhancements is a novel non-pharmacological intervention both for prevention and treatment of sleep deficiency in persons with OA

SUMMARY:
More than 50% of older persons with osteoarthritis (OA) experience disrupted sleep and insomnia symptoms of difficulty falling asleep, awakening during the night, and awakening too early and being unable to fall back to sleep. Because OA pain has been implicated in sleep problems and because physical exercise interventions have been found to improve pain and sleep quality, staying physically active during the daytime is likely advantageous in terms of improving sleep. Physical exercise interventions with a duration between 10 and 16 weeks have been shown to improve quality of sleep in older adults with self-reported disrupted sleep. Unfortunately, recent reports show that older adults with OA are mainly sedentary and few meet national guidelines for recommended amounts of daily physical activity. A self-management intervention that integrates use of mobile technology to prompt older adults to be physically active, provides ongoing monitoring of the amount of their physical activity and includes self-efficacy enhancements is a novel non-pharmacological intervention both for prevention and treatment of sleep deficiency in persons with OA.

The proposed study will involve delivery of automatic physical activity-focused text messages, a novel sleep self-management diary (SleepTight) and motivational interviewing in participants with OA of the hip or knee (most commonly affected joints). The purpose of this Project is to pilot test a new self-management program: MobMPATI, a multidimensional, tailored intervention for sleep deficiency in for older adults with OA. The specific aims are to:

1. Test the acceptability of MobMPATI for older adults with OA and poor sleep quality as a manifestation of sleep deficiency.
2. Test the feasibility of implementing MobMPATI for older adults with OA, as well as collecting electronic data from the sample.
3. Explore pre/posttest changes in self-efficacy, motivation and sleep deficiency measures [total sleep time (TST) and sleep efficiency (SE)] with the MobMPATI intervention.

This study will provide feasibility/acceptability and preliminary data necessary for a larger clinical trial of MobMPATI intervention to encourage physical activity and reduce sedentary behavior in older adults with OA as a way of reducing sleep deficiency. Preliminary testing of the intervention will indicate what measures are more sensitive in promoting self-efficacy and motivation so that a smaller number of outcomes could be monitored to reduce participant burden. This study is the first step in this innovative program of research. The knowledge gained will provide data on the benefit of a potentially cost-effective intervention that could be implemented on a large scale to improve health of older adults with OA.

ELIGIBILITY:
Inclusion Criteria:

>65 years of age

Clinically diagnosed OA of hip or knee

Positive for sleep deficiency, defined as Insomnia Severity Index>=12

Low physical activity based on Rapid Assessment of Physical Activity <=2

Stable use of pain, sleep and/or mood regulating medications over the past month

Resides in Seattle metropolitan area

Exclusion Criteria:

Acute injury associated with hip or knee pain

Inability to stand up without assistance

Memory Impairment Screen for Telephone (MIS-T) score of <4, suggesting cognitive impairment

Severe hearing or visual impairment

An acute episode or change in the treatment of psychiatric problems within the past 3 months

Diagnosed sleep disorder (e.g., sleep disordered breathing; insomnia).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oleg Zaslavsky, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Motivational Interview and Text Messages
Started | 24
Completed | 22
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Motivational Interview and Text Messages
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Mixed Effect Model Inferential Estimates of Longitudinal Changes Across 3 Time Points (Baseline, Week 14, Week 19) in Insomnia Severity Index
Description: Insomnia Severity Index (ISS)
  Score range 0 to 28 at each time point, with higher scores indicating more severe insomnia symptoms
  A single value for change in ISS across three-time points was calculated using linear mixed effect modeling
Time Frame: Assessed at Baseline, week 14, week 19; change from baseline throughout three time points reported
Population: Mixed effect models were utilized because of the time repeated structure of the data. Data collection occasions were also entered in the models to account for change over time. The adjusted for age and gender main effects for time for the ISS was tested for significance and reported as estimates and 95% confidence intervals (CI)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Motivational Interview and Text Messages
Number analyzed (Participants) | 24
units on a scale | -1.24 [-2.43 to -0.05]

2. Primary Outcome: Mixed Effect Model Inferential Estimates of Longitudinal Changes Across Three Time Points (Baseline, Week 14, Week 19) in Actigraphy Total Sleep Time (TST)
Description: Actigraphy Total Sleep Time (TST) in minutes was calculated using baseline, week 14, and week 19 data from a wrist-worn actigraph
  A single value for change in TST across three-time points was calculated using linear mixed effect modeling
  A negative change score indicates lower TST ( in min) over time
Time Frame: Assessed at Baseline, week 14, week 19; change from baseline throughout three time points reported
Population: Mixed effect models were utilized because of the time repeated structure of the data. Data collection occasions were also entered in the models to account for change over time. The adjusted for age and gender main effects for time for the TST was tested for significance and reported as estimates and 95% confidence intervals (CI)
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Motivational Interview and Text Messages
Number analyzed (Participants) | 24
minutes | -4.5 [-13.4 to 4.4]

3. Secondary Outcome: Mixed Effect Model Inferential Estimates of Longitudinal Changes Across Three Time-points (Baseline, Week 14, Week 19) in Self-Efficacy (SE) to Manage Chronic Disease Scale
Description: Self-Efficacy to Manage Chronic Disease Scale
  Score range 1 to 10, with higher scores indicating better efficacy.
  A single value for change in SE across three-time points was calculated using linear mixed effect modeling
  Positive change score indicates an improvement in self-efficacy over time
Time Frame: Assessed at Baseline, week 14, week 19; change from baseline throughout three time points reported
Population: Mixed effect models were utilized because of the time repeated structure of the data. Data collection occasions were also entered in the models to account for change over time. The adjusted for age and gender main effects for time for the self-efficacy was tested for significance and reported as estimates and 95% confidence intervals (CI)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Motivational Interview and Text Messages
Number analyzed (Participants) | 24
score on a scale | 0.28 [-0.07 to 0.63]

4. Secondary Outcome: Mixed Effect Model Inferential Estimates of Longitudinal Changes Across Three Time-points (Baseline, Week 14, Week 19) in Pain Score
Description: Pain
  Score range 1 to 10, with higher scores indicating worse symptoms.
  A single value for change in pain across three-time points was calculated using linear mixed effect modeling
  Positive change score indicates worsening in pain over time
Time Frame: Assessed at Baseline, week 14, week 19; change from baseline throughout three time points reported
Population: Mixed effect models were utilized because of the time repeated structure of the data. Data collection occasions were also entered in the models to account for change over time. The adjusted for age and gender main effects for time for the pain scores was tested for significance and reported as estimates and 95% confidence intervals (CI)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Motivational Interview and Text Messages
Number analyzed (Participants) | 24
score on a scale | -0.13 [-0.47 to 0.20]

5. Secondary Outcome: Mixed Effect Model Inferential Estimates of Longitudinal Changes Across Three Time-points (Baseline, Week 14, Week 19) in Objectively Measured Step Count
Description: Fitbit devices were used to measure weekly step count at baseline, and week 14, and week 19
  A single value for change in step count across three-time points was calculated using linear mixed effect modeling
  A positive change indicates increased step count over time
Time Frame: Assessed at Baseline, week 14, week 19; change from baseline throughout three time points reported
Population: Mixed effect models were utilized because of the time repeated structure of the data. Data collection occasions were also entered in the models to account for change over time. The adjusted for age and gender main effects for time for the step count was tested for significance and reported as estimates and 95% confidence intervals (CI)
Measure: Mean (95% Confidence Interval); unit: step count
Arm/Group | Motivational Interview and Text Messages
Number analyzed (Participants) | 24
step count | 45.6 [-311.6 to 402.9]

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | Motivational Interview and Text Messages
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-18): https://cdn.clinicaltrials.gov/large-docs/87/NCT03160287/Prot_SAP_000.pdf